CLINICAL TRIAL: NCT07264010
Title: Sorafenib Combined With Venetoclax as Pre-emptive Therapy Strategy for Measurable Residual Disease Persisting Acute Myeloid Leukemia: a Prospective, Single-arm, Multicenter Clinical Study
Brief Title: Sorafenib Combined With Venetoclax as Pre-emptive Therapy Strategy for MRD+ AML: a Prospective, Single-arm, Multicenter Clinical Study
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NFEC-2025-434
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukaemia (AML); Measurable Residual Disease (MRD)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual | interventions — Sorafenib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SORA+VEN (Experimental): sorafenib combined with venetoclax
  Interventions: Drug: Sorafenib (SORA); Drug: Venetoclax (VEN)

INTERVENTIONS:
Drug: Sorafenib (SORA) — Sorafenib (SORA) was administered at 400mg twice daily on days 1 to 28.
Drug: Venetoclax (VEN) — Venetoclax (VEN) was administered at 400mg/day on days 1 to 28.

SUMMARY:
The purpose of this study is to explore the efficacy and safety of sorafenib combined with venetoclax as pre-emptive therapy strategy for measurable residual disease persisting acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signing of informed consent form;
* Liver and kidney function: Blood bilirubin ≤ 35 μ mol/L, AST/ALT < 2 times the upper limit of normal, blood creatinine ≤ 150 μ mol/L;
* Normal heart function (EF ≥ 50%, NYHA I/II);
* Physical condition score 0-2 (ECOG score);
* Non pregnant and lactating women. For all women of childbearing age, a pregnancy test must be conducted to determine hCG levels in order to exclude pregnancy status;
* For all men of childbearing age, contraceptive measures must be taken during sorafenib treatment until 3 months after discontinuation.

Exclusion Criteria:

* Acute promyelocytic leukemia;
* Hematological non-remisssion or recurrence;
* Uncontrolled infection or grade 3-4 graft-versus-host disease (GVHD);
* Allergies or contraindications to any of the drugs involved in the protocol;
* Severe organ dysfunction such as heart, liver, kidneys, lungs, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Molecular response rate after three courses of treatment | 1 year
  After three courses of treatment, MRD level decreased ≥1 log10 compared with the pre-treatment

SECONDARY OUTCOMES:
MRD negative rates after three courses of treatment | 1 year
  MRD negative rates after three courses of treatment
Cumulative incidence of relapse (CIR) | 3 year
  Will calculate time from hematological complete rate until relapse.
Event-free survival (EFS) | 3 year
  Will calculate time from assignment until relapse or disease progression.
Overall survival (OS) | 3 year
  Will calculate time from assignment until death from any cause.
Adverse events (AEs) | 3 year
  Treatment-related AEs were defined as those that occurred from the first dose until 30 days after the discontinuation of treatment. The severity of AEs was graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0, except for haematoloical adverse events. Grade 4 hematological adverse events were defined as either an absolute neutrophil count less than 0.5×10⁹cells per L or a platelet count less than 20×10⁹per L.

IPD SHARING:
Plan to Share IPD: No